CLINICAL TRIAL: NCT02374320
Title: Chemical Sympathectomy Following Peripheral Nerve Block With Liposomal Bupivacaine
Brief Title: Exparel as a Nerve Block for Severe Hand Pain
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Jose Soberon, MD (Other)
Responsible Party: Sponsor-Investigator, Jose Soberon, MD, Anesthesiologist, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014.155.C
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: CREST Syndrome; Peripheral Vascular Disease; Raynaud Disease; Scleroderma, Diffuse
MeSH Terms: conditions — CREST Syndrome; Peripheral Vascular Diseases; Raynaud Disease; Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exparel (Experimental): 20 mL liposomal bupivacaine injected once
  Interventions: Drug: liposomal bupivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine — injected as an axillary block

SUMMARY:
The purpose of this study is to investigate whether the use of the study drug (Exparel) is safe and effective for treating circulation problems and pain in the hand or fingers.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status I-IV

Exclusion Criteria:

* True Allergy, not sensitivity to: local anesthetics, midazolam, fentanyl, propofol, ketamine
* Previous surgery or significant trauma involving the radial or ulnar arteries (previous history of angiography and intravascular catheter placement are permitted)
* Pregnancy
* Severe hepatic impairment
* Evidence of infection at or near the proposed needle insertion site
* Any sensorimotor deficit of the ipsilateral upper extremity, whether acute or chronic as determined by the PI and/or designee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Soberon, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exparel (Bupivacaine Liposome Injectable Suspension): 20 mL Exparel (bupivacaine liposome injectable suspension) injected once
  liposomal bupivacaine: injected as an axillary block
Period: Overall Study
Arm/Group | Exparel (Bupivacaine Liposome Injectable Suspension)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exparel
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Radial and Ulnar Arterial Diameter
Description: Radial and ulnar artery diameter was measured at baseline and 60 min after with a Doppler ultrasound system. A marker was used to indicate the site of initial transducer placement on the forearm to ensure that subsequent scans were performed at the same location.
Time Frame: 1 hour
Measure: Mean (Full Range); unit: centimeters
Groups:
- Pre-block (Baseline): 20 mL liposomal bupivacaine injected once
  liposomal bupivacaine: injected as an axillary block
Arm/Group | Pre-block (Baseline) | One Hour Post Block
Number analyzed (Participants) | 13 | 13
centimeters
  Ulnar artery diameter | 0.16 [0.07 to 0.234] | .20 [0.107 to 0.254]
  Radial artery diameter | 0.19 [0.15 to 0.234] | 0.23 [0.15 to 0.336]

2. Secondary Outcome: Pain Measured by Numerical Rating Scale
Description: Numerical rating scale pain scores range from 0 (absence of pain) to 10 (worst pain imaginable)
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Baseline Mean Numerical Rating Scale Pain Score: 20 mL liposomal bupivacaine injected once
  liposomal bupivacaine: injected as an axillary block
Arm/Group | Baseline Mean Numerical Rating Scale Pain Score | Mean Numerical Rating Scale Pain Score at 30 Days
Number analyzed (Participants) | 13 | 13
units on a scale | 6.0 [2 to 10] | 5.2 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Exparel
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes